CLINICAL TRIAL: NCT06286826
Title: Observational Study of Patients Undergoing Surgical Treatment for Oesophageal Atresia: Comparison Between Posterolateral Thoracotomy and Axillary Muscle-sparing Minithoracotomy
Brief Title: A Study of Patients Undergoing Surgical Treatment for Oesophageal Atresia
Status: Recruiting | Type: Observational
Sponsor: Meyer Children's Hospital IRCCS (Other)
Responsible Party: Principal Investigator, Elisa Severi, Principal Investigator, Meyer Children's Hospital IRCCS
Other Study IDs: ATRESO
Record Dates: First submitted 2024-02-19; First posted 2024-02-29 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Atresia Esophagus
MeSH Terms: conditions — Esophageal Atresia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with oesophageal atresia minithoracotomy: Patients with oesophageal atresia who underwent a minithoracotomy between 2011-2021
  Interventions: Procedure: Minithoracotomy
- Patients with oesophageal atresia postero-lateral thoracotomy: Patients with oesophageal atresia who underwent a postero-lateral thoracotomy between 2011-2021
  Interventions: Procedure: Postero-lateral thoracotomy

INTERVENTIONS:
Procedure: Postero-lateral thoracotomy — this incision extends from the anterior axillary line, goes posteriorly behind the scapula and includes the division of the fibres of the latissimus dorsi muscle and the serratus anterior muscle. The latter approach presents the risk of numerous long-term musculoskeletal complications such as costal abnormalities (costal hypoplasia, costal fusion), winged scapula, scoliotic spine posture
  Groups: Patients with oesophageal atresia postero-lateral thoracotomy
Procedure: Minithoracotomy — Minithoracotomy aims to preserve the muscles of the rib cage by retracting or disconnecting them rather than sectioning them (muscle sparing technique)
  Groups: Patients with oesophageal atresia minithoracotomy

SUMMARY:
Oesophageal atresia (EA) is a rare congenital anomaly whose prevalence varies between 1 and 2 per 5000 live births in Europe. This condition is characterised by an interruption of the oesophagus often associated with the presence of a tracheo-oesophageal fistula (FTE).

Although considerable progress has been made in the treatment of AE in recent years, the aetiology of this defect is still not fully understood and several theories have been put forward to explain this phenomenon. What they have in common is an abnormal separation of the primary oesophagus and trachea. The main goal of AE treatment is the closure of the FTE using surgical techniques.

This is a non-profit, multicentre longitudinal observational cohort study. This study will enrol patients who underwent surgery for oesophageal atresia during the period 2011-2021 and are still in follow-up at participating clinical centres.

The primary objective is to assess the incidence of musculoskeletal abnormalities, of any type, in the long term (4 years after surgery) in patients with oesophageal atresia treated surgically by two different approaches: postero-lateral thoracotomy and mini-thoracotomy with muscle preservation

ELIGIBILITY:
Inclusion Criteria:

* Patients with oesophageal atresia (type III according to Ladd's classification);
* Patients who underwent their first operation for oesophageal atresia in the period 2011-2021
* Signature of written informed consent and consent to the study and privacy.

Exclusion Criteria:

* Not signature of written informed consent and consent to the study and privacy.

Ages: 1 Day to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients with oesophageal atresia (type III according to Ladd's classification).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-10-12 (Actual); Primary Completion 2024-10-12 (Estimated); Study Completion 2026-01-12 (Estimated)

PRIMARY OUTCOMES:
incidence of musculoskeletal abnormalities patients with oesophageal atresia treated surgically | Four years after the beginning of the study
  evaluate the incidence of musculoskeletal abnormalities, of all types, in the long term (4 years after surgery) in patients with oesophageal atresia treated surgically using two different approaches: postero-lateral thoracotomy and mini-thoracotomy with muscle preservation.

SECONDARY OUTCOMES:
incidence of musculoskeletal abnormalities in the short term | Six months after surgery
  assess the incidence of musculoskeletal abnormalities in the short term (6 months after surgery);
incidence of musculoskeletal abnormalities in the medium term | Twentyfour months after surgery
  to assess the incidence of musculo-skeletal abnormalities in the medium term (24 months after surgery);
Evaluation of severity of outcomes in the medium, short and long term | One year after the Beginning of the study
  evaluate the severity of outcomes (musculoskeletal abnormalities, respiratory pathologies, eating disorders) in the medium, short and long term. Musculoskeletal abnormalities will be evaluated using the "Trunk Aesthetic Clinical Evaluation (TRACE) Scale"; this scale involves evaluation of shoulder asimmetry (1-3), scapulae asimmetry (1-2), hemi-thorax asimmetry (1-2), waist asimmetry (1-4). Respiratory pathologies are defined as the presence or absence of asthma and recurrent respiratory infections that requires hospitalization (>3 per years). Eating disorders will be defined on the base of the consistence and the dimension of the pieces of food eaten by the child.
Predective Facotrs evaluation | One year after the Beginning of the study
  evaluate the effect of potential predictive factors (such as incision type, intercostal space opening, pleural approach) on abnormalities at different time-points. Musculoskeletal abnormalities will be evaluated using the "Trunk Aesthetic Clinical Evaluation (TRACE) Scale"; this scale involves evaluation of shoulder asimmetry (1-3), scapulae asimmetry (1-2), hemi-thorax asimmetry (1-2), waist asimmetry (1-4).

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Severi, Principal Investigator — Meyer Children's Hospital IRCCS
Locations (3):
- Italy (3):
  - Spedali Civili di Brescia, Brescia
  - Meyer Children's Hospital IRCCS, Florence
  - Ospedale Bambino Gesù di Roma, Roma